CLINICAL TRIAL: NCT02566317
Title: Stand & Move at Work: A Group Randomized Trial
Brief Title: Stand & Move at Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA198971 (NIH)
Record Dates: First submitted 2015-09-22; First posted 2015-10-02 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Hypertension; Diabetes
MeSH Terms: conditions — Obesity; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Move (Active Comparator): A multi-level individual, social, environmental, and organizational intervention targeting increases in light-intensity physical activity in the workplace.
  Interventions: Behavioral: Move
- Stand & Move (Experimental): Move intervention (A multi-level individual, social, environmental, and organizational intervention targeting increases in light-intensity physical activity in the workplace) plus the installation of a sit-stand workstation.
  Interventions: Device: Sit-Stand workstation; Behavioral: Move

INTERVENTIONS:
Device: Sit-Stand workstation — Installation of a sit-stand desk at work
  Arms: Stand & Move
Behavioral: Move — A multi-level individual, social, environmental, and organizational intervention targeting increases in light-intensity physical activity in the workplace

SUMMARY:
A trial testing the efficacy of sit-stand workstations on decreasing sitting time and increasing light-intensity physical activity in samples of office worksites.

DETAILED DESCRIPTION:
With traditional approaches to increasing MVPA (moderate to vigorous physical activity) in the workplace being unsustainable due to the requirement of deliberate and dedicated time away from work, this group-randomized trial will test the efficacy of sit-stand workstations on decreasing sitting time and increasing light-intensity physical activity (LPA) in a highly generalizable sample of office worksites using a multi-level intervention with high potential for dissemination.

ELIGIBILITY:
Inclusion Criteria:

Worksite-level inclusion criteria:

* Size: Small to moderate size worksite (20-60 employees)
* Schedule: >80% of employees full time
* Occupation: Seated office work, primarily computer- and- telephone-based work, little movement or walking
* Wellness environment: Not currently undergoing a wellness program aimed at increasing activity at work
* Workstations: Willing to have sit-stand workstations installed at a worksite
* Willing to be randomized: Willing to be randomized to either intervention conditions

Member-level inclusion criteria:

* Age: 18 years and older
* Health status: Generally good health and able to safely increase LPA and reduce sitting time
* Employment status: Any sedentary job, sitting most of the say, little standing or walking
* Occupation: Traditional sitting desk, willing to have a sit-stand workstation installed at desk
* Workstation: traditional sitting desk;willing to have a sit-stand workstation installed at desk

Exclusion Criteria:

* contraindication to prolonged standing at work

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Buman, PhD, Principal Investigator — Arizona State University; Mark A Pereira, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leonard KS, Larouche M, Mitchell NR, Rydell SA, Toledo MJ, Mullane SL, Hasanaj K, de Brito JN, Buman MP, Pereira MA. Maintenance effects of a multilevel workplace intervention to reduce sedentary time: twenty-four-month follow-up of the group randomized clinical trial 'Stand and Move at Work'. Int J Behav Nutr Phys Act. 2025 Apr 7;22(1):39. doi: 10.1186/s12966-025-01731-w. PMID 40197229
- [Derived] Leonard KS, Mullane SL, Golden CA, Rydell SA, Mitchell NR, Koskan A, Estabrooks PA, Pereira MA, Buman MP. Qualitative comparative analysis of the implementation fidelity of a workplace sedentary reduction intervention. BMC Public Health. 2022 May 31;22(1):1086. doi: 10.1186/s12889-022-13476-3. PMID 35641923
- [Derived] Pereira MA, Mullane SL, Toledo MJL, Larouche ML, Rydell SA, Vuong B, Feltes LH, Mitchell NR, de Brito JN, Hasanaj K, Carlson NG, Gaesser GA, Crespo NC, Oakes JM, Buman MP. Efficacy of the 'Stand and Move at Work' multicomponent workplace intervention to reduce sedentary time and improve cardiometabolic risk: a group randomized clinical trial. Int J Behav Nutr Phys Act. 2020 Oct 27;17(1):133. doi: 10.1186/s12966-020-01033-3. PMID 33109190
- [Derived] Mullane SL, Toledo MJL, Rydell SA, Feltes LH, Vuong B, Crespo NC, Pereira MA, Buman MP. Social ecological correlates of workplace sedentary behavior. Int J Behav Nutr Phys Act. 2017 Aug 31;14(1):117. doi: 10.1186/s12966-017-0576-x. PMID 28859679
- [Derived] Buman MP, Mullane SL, Toledo MJ, Rydell SA, Gaesser GA, Crespo NC, Hannan P, Feltes L, Vuong B, Pereira MA. An intervention to reduce sitting and increase light-intensity physical activity at work: Design and rationale of the 'Stand & Move at Work' group randomized trial. Contemp Clin Trials. 2017 Feb;53:11-19. doi: 10.1016/j.cct.2016.12.008. Epub 2016 Dec 7. PMID 27940181

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Worksites
Groups:
- MOVE+: A multi-level individual, social, environmental, and organizational intervention targeting increases in light-intensity physical activity in the workplace.
  Move: A multi-level individual, social, environmental, and organizational intervention targeting increases in light-intensity physical activity in the workplace
- STAND+: Move intervention (A multi-level individual, social, environmental, and organizational intervention targeting increases in light-intensity physical activity in the workplace) plus the installation of a sit-stand workstation.
  Sit-Stand workstation: Installation of a sit-stand desk at work
  Move: A multi-level individual, social, environmental, and organizational intervention targeting increases in light-intensity physical activity in the workplace
Period: Overall Study
Arm/Group | MOVE+ | STAND+
Started | 276; 12 Worksites | 354; 12 Worksites
Completed | 247; 12 Worksites | 292; 12 Worksites
Not Completed | 29; 0 Worksites | 62; 0 Worksites

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOVE+ | STAND+ | Total
Number analyzed (Participants) | 276 | 354 | 630
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 276 | 354 | 630
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 47 (11) | 45 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 296 | 469
  Male | 103 | 58 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 250 | 239 | 489
  Hispanic | 30 | 57 | 87
  Non-Hispanic Black | 6 | 20 | 26
  Non-Hispanic Asian | 17 | 15 | 32
  Other/Multiracial/Unknown | 18 | 23 | 41
Region of Enrollment [Number; unit: participants]
  United States | 276 | 354 | 630

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Light-intensity Physical Activity at Work From Baseline to 12 Months
Description: Measured via 7d of activPAL accelerometry (value at 12 months minus value at baseline)
Time Frame: 1 year
Population: Among those who completed the study in the MOVE+ arm (n=247), 16 did not have sufficient valid workdays and 7 were missing covariates. Among those who completed the study in the STAND+ arm (n=292), 17 did not have sufficient valid workdays and 12 were missing covariates.
Measure: Mean (95% Confidence Interval); unit: Mean change, minutes per 8hr workday
Arm/Group | MOVE+ | STAND+
Number analyzed (Participants) | 224 | 263
Mean change, minutes per 8hr workday | -0.2 [-2.4 to 2.1] | 2.0 [-0.1 to 4.2]

2. Primary Outcome: Mean Change in Sitting Time at Work From Baseline to 12 Months
Description: Measured via 7d of activPAL accelerometry (value at 12 months minus value at baseline)
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Mean Change, minutes per 8h workday
Arm/Group | MOVE+ | STAND+
Number analyzed (Participants) | 224 | 263
Mean Change, minutes per 8h workday | 6.8 [-4.3 to 17.8] | -52.4 [-62.9 to -42.0]

3. Secondary Outcome: Clustered Metabolic Risk Score From Baseline to 12 Months
Description: Clustered metabolic risk score (fasting glucose, insulin, triglycerides, HDL-cholesterol, blood pressure); value at 12 months minus value at baseline; higher scores indicate better outcome. The Z-score for each component (fasting glucose, insulin, triglycerides, HDL-cholesterol, blood pressure) based on the baseline mean and standard deviation of the entire group was computed and summed for each participant (HDL z-score was subtracted rather than added). The sum of these z-scores represents the metabolic risk score.
Time Frame: 1 year
Population: In MOVE+ (n=247), 10 did not attend posttest visit, 3 were unable to perform a blood draw, 19 refused blood draw, 3 had an insufficent sample, and 8 were missing covariates. In STAND+ (n=292), 16 did not attend posttest visit, 3 were unable to perform a blood draw, 27 refused blood draw, 3 had an insufficent sample, and 5 were missing covariates.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MOVE+ | STAND+
Number analyzed (Participants) | 204 | 238
units on a scale | 0.02 [-0.12 to 0.17] | -0.15 [-0.27 to -0.04]

4. Other Pre Specified Outcome: Sleep Substudy
Description: 24h wrist accelerometry in individuals with minor-moderate sleep complaints
Time Frame: 1 year
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Ambulatory Blood Pressure
Description: Dynamic changes in ambulatory blood pressure in prehypertensives
Time Frame: 3 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Ecological Momentary Assessment of Mood
Description: Periodic monitoring of mood, energy, fatigue in smartphone users
Time Frame: 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Dynamic Glucose Control
Description: Continuous glucose monitoring in prediabetics
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 12 months.
Arm/Group | MOVE+ | STAND+
All-Cause Mortality (participants affected / at risk) | 0/276 | 0/354
Serious Adverse Events (participants affected / at risk) | 0/276 | 0/354
Other Adverse Events (participants affected / at risk) | 0/276 | 0/354

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT02566317/Prot_SAP_000.pdf